CLINICAL TRIAL: NCT05183724
Title: Effects of Radiotherapy and Chemotherapy on Ovarian Function and Post-treatment Pregnancy Outcomes in Women With Nasopharyngeal Carcinoma
Brief Title: Ovarian Function of Nasopharyngeal Carcinoma Women Survivors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Chief Physician, Sun Yat-sen University
Other Study IDs: Ovarian Function of NPC
Record Dates: First submitted 2019-02-16; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; ovarian function; Pregnancy outcomes
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational cohort study aimed to explore the fertility concerns, fertility preservation strategies, fertility status (pregnancy and Ovarian Failure) and birth outcome among young woman Nasopharyngeal carcinoma patients.

DETAILED DESCRIPTION:
The purpose of this study was to explore the effects of radiotherapy and chemotherapy on ovarian function and pregnancy outcome after treatment in female survivors of non-metastatic nasopharyngeal carcinoma, so as to clarify the relationship between ovarian dysfunction after treatment and pregnancy outcome, as well as clarify the relationship between pregnancy after treatment and tumour progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, including WHO II or III ,with no distant metastasis
2. Age between 18-45, female
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal (ULN),serum total bilirubin (TBIL) ≤2.0 times the upper limit of normal (ULN) .
5. Adequate renal function: creatinine clearance rate≥60 ml/min or Creatinine ≤1.5× upper limit of normal value.
6. No history of infertility.
7. No history of hysterectomy or bilateral ovariectomy.
8. Patient have signed on the informed consent, and well understood the objective and procedure of this study

Exclusion Criteria:

1. Histologically or cytologically confirmed with keratinizing squamous cell carcinoma of the nasopharynx.
2. Women in the period of pregnancy, lactation, or reproductive without effective contraceptive measures.
3. Known history of other malignancies (except cured basal cell carcinoma or carcinoma in situ of the cervix).
4. Patients with severe dysfunction of heart, liver, lung, kidney or marrow.
5. Patients with severe, uncontrolled disease or infections.
6. Refuse or fail to sign the informed consent .
7. Patients with personality or mental disorders, incapacity or limited capacity for civil conduct.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Female NPC patients (18 to 45 years old)
Sampling Method: Non-Probability Sample
Enrollment: 602 (Estimated)
Dates: Start 2022-01-10 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Premature Ovarian Failure (POF) | 3 years after Radiotherapy
  Premature Ovarian Failure (POF) was defined as menopause before age 40 years. Menopause was defined as cessation of menstruation at least 1 year before the date of the survey in the absence of pregnancy, breastfeeding, continuous use of progestagens or other medication causing amenorrhea, or surgical removal of uterus and/ or ovaries.

SECONDARY OUTCOMES:
Progress-Free Survival (PFS) | 3 years after Radiotherapy
  Progress-free survival is calculated from the date of registration to the date of the first progress at any site.
Pregnancy and birth outcome | Within 6 month of diagnosis, or 3-5years after Radiotherapy
  The pregnancy history and pregnancy outcome of female Nasopharyngeal carcinoma (NPC) patients before diagnosis of NPC would be investigate Within 6 months of diagnosis.
  The pregnancy events and birth outcome of female NPC patients after diagnosis of NPC would be investigate among 3 to 5years after Radiotherapy.
Overall Survival (OS) | 3 years after Radiotherapy
  The Overall Survival (OS) was defined as the duration from the date of registration assignment to the date of death from any cause or censored at the date of the last follow-up.
Locoregional Relapse-Free Survival (LRFS) | 3 years after Radiotherapy
  The Locoregional Relapse-Free Survival (LRFS) is evaluated and calculated from the date of registration until the day of first locoregional relapse or until the date of the last follow-up visit
Distant Metastasis-Free Survival (DMFS) | 3 years after Radiotherapy
  The DMFS is evaluated and calculated from the date of registration until the day of first distant metastases or until the date of the last follow-up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China